CLINICAL TRIAL: NCT04007419
Title: Promotoras de Donación: Leveraging Community Health Workers to Increase Donor Registration of Older Hispanics
Brief Title: Health Promoters and Organ Donation
Acronym: PdD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R39OT29878
Record Dates: First submitted 2019-06-11; First posted 2019-07-05 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Organ Donation; Donor Designation/Registration
Keywords: Organ donation; Donor designation/registration; Train-the-trainer; Promotora; Community health worker; Lay health educator; Program development; Program evaluation
MeSH Terms: interventions — Tissue and Organ Procurement

STUDY DESIGN:
Intervention Model Description: The study includes focus group interviews with mature Latina and Promotora to inform the development of a web-based educational and communication intervention, as well as an evaluation of the intervention using a nonrandomized, quasi-experimental pragmatic design, pre-post only with no control group to test the impact of the eLearning module on lay health educators' knowledge of organ donation and confidence holding discussions about and promoting organ donation. Additionally, we will examine the impact of the Promotoras de Donación intervention, which will engage trained lay health educators to lead small group sessions with mature Latina, on the women's attitudes about organ donation and donor registration, and rates of donor registration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): The Promotoras de Donación eLearning module will be launched and 40 participating lay health educators trained. Access to the module will be provided via a link to the website embedded in an announcement email. To assess the impact of the Promotoras de Donación eLearning module on lay health educators' knowledge of organ donation and the need for Hispanic donors, and confidence communicating about donation and promoting the act of donor registration, participating lay health educators will complete a brief online survey upon enrollment (pre) and after completing the module (post). Then, trained lay health educators will hold at least 2 small group sessions with mature Latina (6-8 per session); in all, 80 sessions are anticipated with 480 to 640 mature Latina. Participating mature Latina will complete anonymous paper-pencil surveys before and after each session to assess changes in attitudes toward organ donation and donor registration and intent to register as posthumous organ donors.
  Interventions: Behavioral: Health Promoters and Organ Donation

INTERVENTIONS:
Behavioral: Health Promoters and Organ Donation — Promotoras de Donación is a highly engaging and interactive online learning experience, that accommodates multiple learning styles by incorporating a variety of pedagogic approaches. The module consists of two components: a didactic educational component and a skills-based communication component. The didactic component provides basic information about organ donation and transplantation and the need for donors in the Hispanic community, and addresses concerns about donation commonly held by older Latina. The skills-based component provides instruction on the key communication skills needed to effectively engage small groups in discussions about organ donation. This component is intended to build communication self-efficacy or confidence opening the discussion about donation, addressing concerns raised by mature and older women participating in the small group sessions, and promoting the act of donor registration using persuasive, but non-coercive language.
  Other Names: Promotoras de Donación (PdD)

SUMMARY:
Older Hispanics (age 50+ years) are disproportionately overrepresented on the transplant waitlist, but underrepresented as deceased donors and transplant recipients. This application proposes the formative research to design and empirically test an eLearning module, Promotoras de Donación, to train community health workers (i.e., Promotoras), who already provide culturally and linguistically sensitive services to their communities, to discuss and promote organ donation with older Hispanic women in 3 geographically distinct communities across the U.S. The proposed intervention leverages the established and evidence-based Promotoras program to increase rates of donor designation within Hispanic communities across the U.S. and reduce disparities in access to transplantation for this population.

DETAILED DESCRIPTION:
Despite consistently positive attitudes toward organ donation, increasing the number of registered organ donors in the US continues to challenge the professional and research communities. Improving rates of donor designation among ethnic minorities is of particular importance given the need to match donated organs to recipients on blood type and human leukocyte antigens - the best matches are found when the donor and recipient are of the same ethnic background. In Hispanic communities, lay health educators (i.e., Promotoras) are trained to promote behaviors that empower and enable constituents to prevent disease, and increase control over and improve their health. In partnership with leadership of four Promotoras organizations in geographically diverse areas of the U.S. (PA, IL, TX) representing the largest subgroups of the Hispanic population, this pilot study proposes to leverage the preexisting network of lay health educators to advocate for organ donation and promote donor registration (first person consent) among female Hispanics over the age of 50. Specifically, this study will collect the formative data needed to design an educational and behavioral communication eLearning module for Promotoras and test the impact of the training on Promotoras' knowledge of organ donation, confidence discussing and promoting donor registration, and efficacy increasing rates of donor registration among mature and older Hispanic women. Focus group interviews with Hispanic women and Promotoras will identify the information needs and concerns about organ donation registration of these two groups; interviews with lay educators will also gauge interactivity preferences as well as content and design issues for the resulting web-based training (Aim 1). These data will be used to develop an eLearning module to educate Promotoras about organ donation and train them to discuss donation and promote donor registration (Aim 2). A brief quantitative survey will assess the impact of the module on knowledge of organ donation and confidence (communication self-efficacy) discussing donation and promoting donor designation. We will evaluate Promotoras' efficacy promoting organ donation by assessing the number of Hispanic women age 50 and over who register as posthumous organ donors as a proportion of all women attending small group sessions led by trained Promotoras (Aim 3). If effective, the eLearning module could easily be disseminated nationally to train Promotoras to discuss and promote organ donation. Ultimately, this 'train-the-trainer' study has the potential to increase rates of donor registration among Hispanic communities in the U.S. and help to reduce disparities in access to transplantation for this population.

ELIGIBILITY:
Inclusion Criteria:

* Lay health educators (Promotora): Lay health educators must be at least 18 years of age, have completed all required Promotoras training, and have actively worked with the local Hispanic community within 3 months of recruitment.
* Mature Latina: Eligible women must be at least 50 years of age, with no obvious cognitive impairment.

Exclusion Criteria:

* Lay health educators (Promotora): Untrained lay health educators or those currently in training at their respective organizations will be deemed ineligible, as will individuals who are not actively working as a Promotora at the time of recruitment/enrollment.
* Mature Latina: Hispanic women under the age of 50, or those with obvious cognitive impairment will be deemed ineligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Donor registration | 3 months
  The proportion of mature Latina attending the trained lay health educator-led small group sessions who also register their intent to become a posthumous organ, tissue and eye donor

SECONDARY OUTCOMES:
Communication self-efficacy | 3 months
  Lay health educators will be asked to rate their level of confidence managing 10 communication skills relevant to discussing organ donation and promoting donor registration along numerical scales ranging from 0 (not at all confident) to 100 (totally confident). A global self-efficacy score will be obtained by summing the ratings for each item.
Knowledge of organ donation | 3 months
  A series of 10 true/false questions previously developed and used to assess knowledge of organ donation in a community sample of Hispanic Americans. A global knowledge score will be created as the sum of all correctly answered questions, ranging from 0 to 10.

OTHER OUTCOMES:
Donation intentions | 3 months
  A single, 4-point Likert-type item will agreement with the following statement: I plan to register as an organ donor in the next month (1-strongly disagree/4-strongly agree). The two categories representing agreement and disagreement, respectively, will be collapsed to create a dichotomous variable indicating intentions to register (1-yes/0-no).
Support for organ donation | 3 months
  We will capture participants' general support for organ donation using a single 5-point Likert type item. The question will ask respondents to indicate the extent to which they support organ donation (1-not at all/5-totally).
Perceptions of the Promotoras de Donación eLearning module | 3 months
  A series of 10, 4-point Likert-type questions will ascertain perceptions of the web-based eLearning module, including organization, length, realism, and interest in the material covered. A single 5-point Likert-type item will capture respondents' rating of the overall quality of the module (1-poor/5-excellent). Finally, two open-ended questions will ask respondents to indicate their most and least liked aspects of the module.

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Gardiner (Traino), PhD, MPH, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available for use by written request to the Principal Investigator. Specifically, focus group and survey data collected from lay health educators and mature Latina will be shared in ways in which participants' privacy and confidentiality are secured. Any identifying information in the data will be redacted before sharing. In an effort to provide further protection from the deductive identification of participants, parties requesting data will be asked to agree to use the data solely for research purposes, to refrain from identifying participants in any manner, to secure the data electronically through encryption and/or password protection, and to return or destroy the data upon completion of the analyses.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study will be available after publication of the study's major findings
Access Criteria: Written request to the Principal Investigator (Heather Gardiner).

REFERENCES:
- [Background] Christmas AB, Mallico EJ, Burris GW, Bogart TA, Norton HJ, Sing RF. A paradigm shift in the approach to families for organ donation: honoring patients' wishes versus request for permission in patients with Department of Motor Vehicles donor designations. J Trauma. 2008 Dec;65(6):1507-9; discussion 1509-10. doi: 10.1097/TA.0b013e31818a5cf0. PMID 19077650
- [Background] Traino HM, Siminoff LA. Attitudes and acceptance of First Person Authorization: a national comparison of donor and nondonor families. J Trauma Acute Care Surg. 2013 Jan;74(1):294-300. doi: 10.1097/TA.0b013e318270dafc. PMID 23147186
- [Background] Siminoff LA, Agyemang AA, Traino HM. Consent to organ donation: a review. Prog Transplant. 2013 Mar;23(1):99-104. doi: 10.7182/pit2013801. PMID 23448829
- [Background] Gallup Organization. The American public's attitudes toward organ donation and transplantation. Boston: The Partnership for Organ Donation; 1993.
- [Background] U.S. Department of Health and Human Services, Health Resources and Services Administration, Healthcare Systems Bureau, 2012 National Survey of Organ Donation Attitudes and Behaviors. Rockville, Maryland: U.S. Department of Health and Human Services, 2013.
- [Background] United States Renal Data System. 2015 USRDS annual data report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2015.
- [Background] Hoerger TJ, Simpson SA, Yarnoff BO, Pavkov ME, Rios Burrows N, Saydah SH, Williams DE, Zhuo X. The future burden of CKD in the United States: a simulation model for the CDC CKD Initiative. Am J Kidney Dis. 2015 Mar;65(3):403-11. doi: 10.1053/j.ajkd.2014.09.023. Epub 2014 Nov 5. PMID 25468386
- [Background] Grams ME, Chow EK, Segev DL, Coresh J. Lifetime incidence of CKD stages 3-5 in the United States. Am J Kidney Dis. 2013 Aug;62(2):245-52. doi: 10.1053/j.ajkd.2013.03.009. Epub 2013 Apr 6. PMID 23566637
- [Background] Eggers PW. Has the incidence of end-stage renal disease in the USA and other countries stabilized? Curr Opin Nephrol Hypertens. 2011 May;20(3):241-5. doi: 10.1097/MNH.0b013e3283454319. PMID 21422925
- [Background] Scaglione S, Kliethermes S, Cao G, Shoham D, Durazo R, Luke A, Volk ML. The Epidemiology of Cirrhosis in the United States: A Population-based Study. J Clin Gastroenterol. 2015 Sep;49(8):690-6. doi: 10.1097/MCG.0000000000000208. PMID 25291348
- [Background] Lim YS, Kim WR. The global impact of hepatic fibrosis and end-stage liver disease. Clin Liver Dis. 2008 Nov;12(4):733-46, vii. doi: 10.1016/j.cld.2008.07.007. PMID 18984463
- [Background] Lazo M, Hernaez R, Eberhardt MS, Bonekamp S, Kamel I, Guallar E, Koteish A, Brancati FL, Clark JM. Prevalence of nonalcoholic fatty liver disease in the United States: the Third National Health and Nutrition Examination Survey, 1988-1994. Am J Epidemiol. 2013 Jul 1;178(1):38-45. doi: 10.1093/aje/kws448. Epub 2013 May 23. PMID 23703888
- [Background] Kim HJ, Lee HW. Important predictor of mortality in patients with end-stage liver disease. Clin Mol Hepatol. 2013 Jun;19(2):105-15. doi: 10.3350/cmh.2013.19.2.105. Epub 2013 Jun 27. PMID 23837134
- [Background] Ahmed A, Keeffe EB. Current indications and contraindications for liver transplantation. Clin Liver Dis. 2007 May;11(2):227-47. doi: 10.1016/j.cld.2007.04.008. PMID 17606204
- [Background] Rein DB, Wittenborn JS, Weinbaum CM, Sabin M, Smith BD, Lesesne SB. Forecasting the morbidity and mortality associated with prevalent cases of pre-cirrhotic chronic hepatitis C in the United States. Dig Liver Dis. 2011 Jan;43(1):66-72. doi: 10.1016/j.dld.2010.05.006. Epub 2010 Jun 17. PMID 20739252
- [Background] Singal AK, Anand BS. Recent trends in the epidemiology of alcoholic liver disease. Clin Liver Dis (Hoboken). 2013 Apr 24;2(2):53-56. doi: 10.1002/cld.168. eCollection 2013 Apr. No abstract available. PMID 30992823
- [Background] Wong RJ, Aguilar M, Cheung R, Perumpail RB, Harrison SA, Younossi ZM, Ahmed A. Nonalcoholic steatohepatitis is the second leading etiology of liver disease among adults awaiting liver transplantation in the United States. Gastroenterology. 2015 Mar;148(3):547-55. doi: 10.1053/j.gastro.2014.11.039. Epub 2014 Nov 25. PMID 25461851
- [Background] Schuppan D, Afdhal NH. Liver cirrhosis. Lancet. 2008 Mar 8;371(9615):838-51. doi: 10.1016/S0140-6736(08)60383-9. PMID 18328931
- [Background] Carrion AF, Ghanta R, Carrasquillo O, Martin P. Chronic liver disease in the Hispanic population of the United States. Clin Gastroenterol Hepatol. 2011 Oct;9(10):834-41; quiz e109-10. doi: 10.1016/j.cgh.2011.04.027. Epub 2011 May 12. PMID 21628000
- [Background] Lazo M, Bilal U, Perez-Escamilla R. Epidemiology of NAFLD and Type 2 Diabetes: Health Disparities Among Persons of Hispanic Origin. Curr Diab Rep. 2015 Dec;15(12):116. doi: 10.1007/s11892-015-0674-6. PMID 26468154
- [Background] Deedat S, Kenten C, Morgan M. What are effective approaches to increasing rates of organ donor registration among ethnic minority populations: a systematic review. BMJ Open. 2013 Dec 20;3(12):e003453. doi: 10.1136/bmjopen-2013-003453. PMID 24362010
- [Background] Breitkopf CR. Attitudes, beliefs and behaviors surrounding organ donation among Hispanic women. Curr Opin Organ Transplant. 2009 Apr;14(2):191-5. doi: 10.1097/mot.0b013e328329255c. PMID 19469039
- [Background] Alvaro EM, Jones SP, Robles AS, Siegel JT. Predictors of organ donation behavior among Hispanic Americans. Prog Transplant. 2005 Jun;15(2):149-56. doi: 10.1177/152692480501500207. PMID 16013463
- [Background] Frates J, Garcia Bohrer G. Hispanic perceptions of organ donation. Prog Transplant. 2002 Sep;12(3):169-75. doi: 10.1177/152692480201200303. PMID 12371041
- [Background] Downing K, Jones LL. Designing an educational strategy for increasing organ donor registration among older adults. Prog Transplant. 2008 Dec;18(4):290-6. doi: 10.1177/152692480801800412. PMID 19186582
- [Background] Quick BL, Anker AE, Feeley TH, Morgan SE. An examination of three theoretical models to explain the organ donation attitude--registration discrepancy among mature adults. Health Commun. 2016;31(3):265-74. doi: 10.1080/10410236.2014.947468. Epub 2015 Aug 25. PMID 26305921
- [Background] Hoyert DL. 75 years of mortality in the United States, 1935-2010. NCHS Data Brief. 2012 Mar;(88):1-8. PMID 22617094
- [Background] Colby SL, Ortman JM. Projections of the size and composition of the U.S. population: 2014 to 2060. Population Estimates and Projections. Current Population Reports. U.S. Census Bureau; 2015.
- [Background] Yracheta JM, Alfonso J, Lanaspa MA, Roncal-Jimenez C, Johnson SB, Sanchez-Lozada LG, Johnson RJ. Hispanic Americans living in the United States and their risk for obesity, diabetes and kidney disease: Genetic and environmental considerations. Postgrad Med. 2015 Jun;127(5):503-10. doi: 10.1080/00325481.2015.1021234. Epub 2015 Mar 7. PMID 25746679
- [Background] Kemmer N, Neff GW. Liver transplantation in the ethnic minority population: challenges and prospects. Dig Dis Sci. 2010 Apr;55(4):883-9. doi: 10.1007/s10620-009-0803-7. Epub 2009 Apr 24. PMID 19390965
- [Background] Dominguez K, Penman-Aguilar A, Chang MH, Moonesinghe R, Castellanos T, Rodriguez-Lainz A, Schieber R; Centers for Disease Control and Prevention (CDC). Vital signs: leading causes of death, prevalence of diseases and risk factors, and use of health services among Hispanics in the United States - 2009-2013. MMWR Morb Mortal Wkly Rep. 2015 May 8;64(17):469-78. PMID 25950254
- [Background] Salim A, Schulman D, Ley EJ, Berry C, Navarro S, Chan LS. Contributing factors for the willingness to donate organs in the Hispanic American population. Arch Surg. 2010 Jul;145(7):684-9. doi: 10.1001/archsurg.2010.110. PMID 20644132
- [Background] Saade M, Morales-Otero L, Davis J, Torres E, Gonzalez Z, Santiago-Delpin EA. A 16-fold increase in organ donation in a Hispanic population. Transplant Proc. 2008 May;40(4):1005-7. doi: 10.1016/j.transproceed.2008.03.120. PMID 18555100
- [Background] Baru JS, Lucas BR, Martinez C, Brauner D. Organ donation among undocumented hispanic immigrants: an assessment of knowledge and attitudes. J Clin Ethics. 2013 Winter;24(4):364-72. PMID 24597424
- [Background] Brown CV, Foulkrod KH, Dworaczyk S, Thompson K, Elliot E, Cooper H, Coopwood B. Barriers to obtaining family consent for potential organ donors. J Trauma. 2010 Feb;68(2):447-51. doi: 10.1097/TA.0b013e3181caab8f. PMID 20154557
- [Background] U.S. Department of Health and Human Services. Report on the Division of Transplantation's Grant Program 1999-2004: Social and Behavioral Interventions to Increase Organ Donation. Institute for Campaign Research and Evaluation. 2005.
- [Background] Salim A, Bery C, Ley EJ, Schulman D, Navarro S, Zheng L, Chan LS. A focused educational program after religious services to improve organ donation in Hispanic Americans. Clin Transplant. 2012 Nov-Dec;26(6):E634-40. doi: 10.1111/ctr.12036. Epub 2012 Oct 29. PMID 23106648
- [Background] Hurtado S. Matrisocialidad Caracas: Edición EBUC=FACES/UCV;1998.
- [Background] U.S. Department of Health and Human Services, Health Resources and Services Administration, Bureau of Health Professions. Community Health Worker National Workforce Study; 2007.
- [Background] Ayala GX, Vaz L, Earp JA, Elder JP, Cherrington A. Outcome effectiveness of the lay health advisor model among Latinos in the United States: an examination by role. Health Educ Res. 2010 Oct;25(5):815-40. doi: 10.1093/her/cyq035. Epub 2010 Jul 5. PMID 20603384
- [Background] University of Arizona. A Summary of the National Community Health Advisor Study. Annie E. Casey Foundation. 1998.
- [Background] Lujan J, Ostwald SK, Ortiz M. Promotora diabetes intervention for Mexican Americans. Diabetes Educ. 2007 Jul-Aug;33(4):660-70. doi: 10.1177/0145721707304080. PMID 17684167
- [Background] McCloskey J. Promotores as partners in a community-based diabetes intervention program targeting Hispanics. Fam Community Health. 2009 Jan-Mar;32(1):48-57. doi: 10.1097/01.FCH.0000342816.87767.e6. PMID 19092434
- [Background] Byrd TL, Wilson KM, Smith JL, Coronado G, Vernon SW, Fernandez-Esquer ME, Thompson B, Ortiz M, Lairson D, Fernandez ME. AMIGAS: a multicity, multicomponent cervical cancer prevention trial among Mexican American women. Cancer. 2013 Apr 1;119(7):1365-72. doi: 10.1002/cncr.27926. Epub 2012 Dec 21. PMID 23280399
- [Background] Fernandez ME, Gonzales A, Tortolero-Luna G, Williams J, Saavedra-Embesi M, Chan W, Vernon SW. Effectiveness of Cultivando la Salud: a breast and cervical cancer screening promotion program for low-income Hispanic women. Am J Public Health. 2009 May;99(5):936-43. doi: 10.2105/AJPH.2008.136713. Epub 2009 Mar 19. PMID 19299678
- [Background] Sosa ET, Biediger-Friedman L, Yin Z. Lessons learned from training of promotores de salud for obesity and diabetes prevention. J Health Dispar Res Prac 6(1): 1, 2013.
- [Background] Staten LK, Cutshaw CA, Davidson C, Reinschmidt K, Stewart R, Roe DJ. Effectiveness of the Pasos Adelante chronic disease prevention and control program in a US-Mexico border community, 2005-2008. Prev Chronic Dis. 2012;9:E08. Epub 2011 Dec 15. PMID 22172175
- [Background] Balcazar H, Alvarado M, Cantu F, Pedregon V, Fulwood R. A promotora de salud model for addressing cardiovascular disease risk factors in the US-Mexico border region. Prev Chronic Dis. 2009 Jan;6(1):A02. Epub 2008 Dec 15. PMID 19080008
- [Background] U.S. Department of Health and Human Services. HHS action plan to reduce racial and ethnic health disparities: A nation free of disparities in health and health care; 2011.
- [Background] Yarber L, Brownson CA, Jacob RR, Baker EA, Jones E, Baumann C, Deshpande AD, Gillespie KN, Scharff DP, Brownson RC. Evaluating a train-the-trainer approach for improving capacity for evidence-based decision making in public health. BMC Health Serv Res. 2015 Dec 12;15:547. doi: 10.1186/s12913-015-1224-2. PMID 26652172
- [Background] Ray ML, Wilson MM, Wandersman A, Meyers DC, Katz J. Using a training-of-trainers approach and proactive technical assistance to bring evidence based programs to scale: an operationalization of the interactive systems framework's support system. Am J Community Psychol. 2012 Dec;50(3-4):415-27. doi: 10.1007/s10464-012-9526-6. PMID 22711269
- [Background] Muramoto ML, Connolly T, Strayer LJ, Ranger-Moore J, Blatt W, Leischow R, Leischow S. Tobacco cessation skills certification in Arizona: application of a state wide, community based model for diffusion of evidence based practice guidelines. Tob Control. 2000 Dec;9(4):408-14. doi: 10.1136/tc.9.4.408. PMID 11106711
- [Background] Orfaly RA, Frances JC, Campbell P, Whittemore B, Joly B, Koh H. Train-the-trainer as an educational model in public health preparedness. J Public Health Manag Pract. 2005 Nov;Suppl:S123-7. doi: 10.1097/00124784-200511001-00021. PMID 16205531
- [Background] Rubak S, Mortensen L, Ringsted C, Malling B. A controlled study of the short- and long-term effects of a Train the Trainers course. Med Educ. 2008 Jul;42(7):693-702. doi: 10.1111/j.1365-2923.2008.03044.x. Epub 2008 May 23. PMID 18507769
- [Background] Greif R, Becker CB, Hildebrandt T. Reducing eating disorder risk factors: A pilot effectiveness trial of a train-the-trainer approach to dissemination and implementation. Int J Eat Disord. 2015 Dec;48(8):1122-31. doi: 10.1002/eat.22442. Epub 2015 Aug 18. PMID 26281792
- [Background] Marsh T, Derose KP, Rios M, Cohen D. Promotoras as data collectors in a large study of physical activity in parks. Health Promot Pract. 2015 May;16(3):354-61. doi: 10.1177/1524839914563076. Epub 2015 Feb 3. PMID 25649234
- [Background] Johnson CM, Sharkey JR, Dean WR, St John JA, Castillo M. Promotoras as research partners to engage health disparity communities. J Acad Nutr Diet. 2013 May;113(5):638-42. doi: 10.1016/j.jand.2012.11.014. Epub 2013 Feb 1. No abstract available. PMID 23375463
- [Background] Sharkey JR, Dean WR, St John JA, Huber JC Jr. Using direct observations on multiple occasions to measure household food availability among low-income Mexicano residents in Texas colonias. BMC Public Health. 2010 Jul 29;10:445. doi: 10.1186/1471-2458-10-445. PMID 20670423
- [Background] O'Hegarty M, Pederson LL, Thorne SL, Caraballo RS, Evans B, Athey L, McMichael J. Customizing survey instruments and data collection to reach Hispanic/Latino adults in border communities in Texas. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S159-64. doi: 10.2105/AJPH.2009.167338. Epub 2010 Feb 10. PMID 20147687
- [Background] Rhodes SD, Foley KL, Zometa CS, Bloom FR. Lay health advisor interventions among Hispanics/Latinos: a qualitative systematic review. Am J Prev Med. 2007 Nov;33(5):418-27. doi: 10.1016/j.amepre.2007.07.023. PMID 17950408
- [Background] Gordon EJ, Feinglass J, Carney P, Vera K, Olivero M, Black A, O'Connor K, MacLean J, Nichols S, Sageshima J, Preczewski L, Caicedo JC. A Culturally Targeted Website for Hispanics/Latinos About Living Kidney Donation and Transplantation: A Randomized Controlled Trial of Increased Knowledge. Transplantation. 2016 May;100(5):1149-60. doi: 10.1097/TP.0000000000000932. PMID 26444846
- [Background] Gordon EJ, Feinglass J, Carney P, Ramirez D, Olivero M, O'Connor K, MacLean J, Brucker J, Caicedo JC. An interactive, bilingual, culturally targeted website about living kidney donation and transplantation for hispanics: development and formative evaluation. JMIR Res Protoc. 2015 Apr 20;4(2):e42. doi: 10.2196/resprot.3838. PMID 25896143
- [Background] Morgan SE, Miller JK. Beyond the organ donor card: the effect of knowledge, attitudes, and values on willingness to communicate about organ donation to family members. Health Commun. 2002;14(1):121-34. doi: 10.1207/S15327027HC1401_6. PMID 11853207
- [Background] Morgan SE, Miller JK. Communicating about gifts of life: the effect of knowledge, attitudes, and altruism on behavior and behavioral intentions regarding organ donation. J Applied Commun Res. 2002; 30:163-78. doi: 10.1080/00909880216580.
- [Background] Crano WD. Vested interest, symbolic politics, and attitude-behavior consistency. J Pers Soc Psychol. 1997 Mar;72(3):485-91. doi: 10.1037//0022-3514.72.3.485. PMID 9120779
- [Background] Crano WD, Prislin R. Components of vested interest and attitude-behavior consistency. Bas Appl Soc Psychol. 1995;17:1-21. doi:10.1080/01973533.1995.9646129.
- [Background] Morgan SE, Miller JK, Arasaratnam LA. Similarities and differences between African Americans' and European Americans' attitudes, knowledge, and willingness to communicate about organ donation. J Applied Soc Psychol. 2003;33:693-715. doi: 10.1111/j.1559-1816.2003.tb01920.x
- [Background] Morgan SE. The power of talk: African Americans' communication with family members about organ donation and its impact on the willingness to donate. J Soc Pers Rel. 2004;21:112-24. doi: 10.1177/0265407504039845
- [Background] Robinson DH, Perryman JP, Thompson NJ, Amaral S, Arriola KR. Testing the utility of a modified organ donation model among African American adults. J Behav Med. 2012 Jun;35(3):364-74. doi: 10.1007/s10865-011-9363-3. Epub 2011 Jun 23. PMID 21698439
- [Background] Anker AE, Feeley TH. Are nonparticipants in prosocial behavior merely innocent bystanders? Health Commun. 2011 Jan;26(1):13-24. doi: 10.1080/10410236.2011.527618. PMID 21308580
- [Background] Anker AE, Feeley TH, Kim H. Examining the attitude-behavior relationship in prosocial donation domains. J Appl Soc Psychol. 2010;40:1293-1324.
- [Background] Krueger RA. Focus groups: A practical guide for applied research, 2nd ed. Thousand Oaks, CA: Sage; 1994.
- [Background] Kamberelis G, Dimitriadis G. Focus groups: contingent articulations of pedagogy, politics, and inquiry. NK Denzin & YS Lincoln. The SAGE Handbook of Qualitative Research. 2011.
- [Background] Asbury J-E. Overview of focus group research. Qual Health Res. 1995;5(4):414-20.
- [Background] Vaughn S, Schumm JS, Sinagub J. Focus group interviews in education and psychology. Thousand Oaks, CA: Sage; 1996.
- [Background] Spitzberg BH, Cupach WR. Interpersonal communication competence. Beverly Hills, CA: Sage; 1984.
- [Background] Hargie O. Handbook of communication skills. New York: Routledge; 2006.
- [Background] Leont'ev AN. The problem of activity in psychology. J Rus East Europ Psychol. 1974;13(2): 4-33.
- [Background] Dewey J. Democracy and education: An introduction to the philosophy of education. The Macmillan Company; 1916.
- [Background] Hannafin MJ. Interaction Strategies and Emerging Instructional Technologies: Psychological Perspectives. Can J Educ Commun. 1989; 18(3): 167-79.
- [Background] Holmberg B. Theory and practice of distance education. London: Routledge; 1989.
- [Background] Stephenson J, Imrie J. Why do we need randomised controlled trials to assess behavioural interventions? BMJ. 1998 Feb 21;316(7131):611-3. doi: 10.1136/bmj.316.7131.611. No abstract available. PMID 9518919
- [Background] Lindquist R, Wyman JF, Talley KM, Findorff MJ, Gross CR. Design of control-group conditions in clinical trials of behavioral interventions. J Nurs Scholarsh. 2007;39(3):214-21. doi: 10.1111/j.1547-5069.2007.00171.x. PMID 17760793
- [Background] Friedman LM, Furberg CD, DeMets DL. Fundamentals of Clinical Trials, 4th ed. New York, NY: Springer; 2010.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Strauss A, Corbin J. Basics of qualitative research: grounded theory procedures and techniques. Newbury Park, CA; Sage; 1990.
- [Background] Berg BL. Qualitative research methods for the social sciences, 6th ed. Boston, MA: Allyn & Bacon; 2007.
- [Background] Mays N, Pope C. Qualitative research in health care. Assessing quality in qualitative research. BMJ. 2000 Jan 1;320(7226):50-2. doi: 10.1136/bmj.320.7226.50. No abstract available. PMID 10617534
- [Background] Neuendorf KA. The content analysis guidebook. Thousand Oaks, CA: Sage; 2002.
- [Derived] Gordon EJ, Gardiner H, Siminoff LA, Kelly PJ, Agu C, Urbanski M, Alolod GP, Benitez A, Hernandez I, Guinansaca N, Ramos Winther L, Bergeron CD, Kim R, Montalvo A, Gonzalez T. Donor Designation Among Mature Latinas and Lay Health Educators (Promotoras): A Mixed-Methods Study. Health Educ Behav. 2021 Dec;48(6):805-817. doi: 10.1177/1090198120976351. Epub 2020 Dec 21. PMID 33345620
- [Derived] Alolod GP, Gardiner H, Agu C, Turner JL, Kelly PJ, Siminoff LA, Gordon EJ, Norden R, Daly TA, Benitez A, Hernandez I, Guinansaca N, Winther LR, Bergeron CD, Montalvo A, Gonzalez T. A Culturally Targeted eLearning Module on Organ Donation (Promotoras de Donacion): Design and Development. J Med Internet Res. 2020 Jan 13;22(1):e15793. doi: 10.2196/15793. PMID 31929102
- See also: Organ Procurement and Transplantation Network. U.S. Department of Health & Human Services. — https://optn.transplant.hrsa.gov/data/view-data-reports/national-data/
- See also: Revised Uniform Anatomical Gift Act (2006). Last Revised or Amended in 2009. National Conference of Commissioners of Uniform State Laws — https://www.uniformlaws.org/committees/community-home?CommunityKey=015e18ad-4806-4dff-b011-8e1ebc0d1d0f
- See also: Donate Life America. 2015 Annual Update — https://donatelife.net/2015-dla-annual-update-released/
- See also: U.S. Census Bureau. U.S. Census Bureau projections show a slower growing, older, more diverse nation a half century from now — https://www.census.gov/newsroom/releases/archives/population/cb12-243.html?cssp=SERP
- See also: U.S. Census Bureau. American Fact Finder — http://factfinder.census.gov
- See also: U.S. Department of Health & Human Services, Office of Minority Health, Think Cultural Health. Promoting Healthy Choices and Community Changes: An E-learning Program for Promotores De Salud — http://promotores.thinkculturalhealth.hhs.gov